CLINICAL TRIAL: NCT03597503
Title: Assessment of Efficacy and Safety of SPN-810 for the Treatment of Impulsive Aggression (IA) in Adolescent Subjects With Attention Deficit/Hyperactivity Disorder (ADHD) in Conjunction With Standard ADHD Treatment
Brief Title: Treatment of Impulsive Aggression (IA) in Adolescent With ADHD in Conjunction With Standard ADHD Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision, not related to safety
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 810P503
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel group, two-arm, placebo-controlled study with flexible dosing
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flexible dose of SPN-810 (Experimental): Subjects treated with flexible dose of SPN-810
  Interventions: Drug: SPN-810
- Placebo (Placebo Comparator): Subjects treated with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-810 — Flexible dose
  Arms: Flexible dose of SPN-810
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the effect of SPN-810 for the treatment of impulsive aggression (IA) in adolescents diagnosed with ADHD when taken in conjunction with standard ADHD treatment.

DETAILED DESCRIPTION:
This study was an addition to the pediatric studies (CHIME 1 and CHIME 2) to assess the efficacy and safety of SPN-810 in the improvement of impulsive aggression (IA) behaviors in adolescents with ADHD.

SPN-810 was administered in patients diagnosed with ADHD and associated features of IA, who were currently treated with an FDA-approved standard ADHD treatment and displayed persistent IA behaviors. The frequency of impulsive aggressive behaviors was assessed as a primary outcome.

.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise, healthy non-smoking, male and females adolescents (12-17 years of age at the time of screening) with a primary diagnosis of ADHD and currently taking an optimized FDA-approved ADHD medication.
* IA confirmed at screening using R-MOAS scale and Vitiello Aggression Questionnaire.

Exclusion Criteria:

* History or current diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia and other psychotic disorders, personality disorder, Tourette's syndrome or dissociative disorder, autism spectrum disorder, pervasive developmental disorder, obsessive compulsive disorder, post-traumatic stress disorder, or intermittent explosive disorder.
* Currently meeting DSM-5 criteria for pervasive developmental disorder, obsessive compulsive disorder, post-traumatic stress disorder or intermittent explosive disorder.
* Known or suspected intelligence quotient (IQ) <70, active suicidal plan/intent or active suicidal thought, criminal arrest, alcohol or drug use or pregnancy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - ProScience, Culver City, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Children's National Medical Center/Children's Research Institute, Washington D.C., District of Columbia
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Meridien Research aka Florida Clinical Research Center, LLC, Lakeland, Florida
  - Florida Clinical Research Center, LLC., Maitland, Florida
  - Miami Clinical Research, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - University of South Florida- Dept. of Psychiatry and Neurosciences, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR Conventions Research, Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Hugo W Moser Research Institute at Kennedy Krieger, Baltimore, Maryland
  - St. Charles Psychiatric Associates Midwest Research Center, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Hassmann Research Institute, Berlin, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - Ohio State University Nisonger Center Clinical Trials Program, Columbus, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - CNS Healthcare, Memphis, Tennessee
  - Texas Physicians Medical Research Group, Arlington, Texas
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - Gaolin Research, LLC, Beaumont, Texas
  - Relaro Medical Trials, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Houston Clinical Trials, Houston, Texas
  - Dicovery MM Services Inc. Houston, Houston, Texas
  - FMCScience, Lampasas, Texas
  - Discovery MM Service, Inc. Missouri, Missouri City, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Ericksen Research & Development, Clinton, Utah
  - Aspen Clinical Research, Orem, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent a 15-day baseline period (up to -Day 15), were randomized on Day 1 to receive either placebo or SPN-180, and then entered a 2- week titration phase followed by a 3-weeks maintenance phase, and then a 1-week taper phase.
Groups:
- Flexible Dose of SPN-810: Subjects treated with flexible dose of SPN-810 (36, 45 or 54 mg/day).
Period: Overall Study
Arm/Group | Placebo | Flexible Dose of SPN-810
Started (Number of subjects is based on the Safety Population, defined as all subjects who received at least 1 dose of study drug and had at least one post-baseline safety assessment.) | 20 | 21
Treated | 20 | 21
Completed | 18 | 17
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Participants is based on the Safety Population, defined as all subjects who received at least 1 dose of study drug and had at least one post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Flexible Dose of SPN-810 | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (1.43) | 13.2 (1.25) | 13.1 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Effect of SPN-810 Treatment on the Frequency of Impulsive Aggression (IA) Behaviors Measured by the Impulsive Aggression Diary
Description: The primary efficacy endpoint was percent change (PCHT) in the frequency (unweighted score) of IA behaviors per 7 days in the treatment (titration and maintenance) period relative to the baseline period calculated over the number of days with non-missing IA diary data. PCHT was then calculated as 100 x (T - B)/B, where T and B are IA behavior frequencies per 7 days during the treatment period (from Day 2 through Visit 7, inclusive) and baseline period (Day ≤1), respectively. The IA behavior frequency per 7 days is defined as (SUM/DAY) x 7, where SUM is the total of the IA behaviors reported in the subject IA diary, and DAY is the number of days with a non-missing IA score in the subject IA diary during the specified study period.
Time Frame: Daily measure from Visit 2 (Day -15) to Visit 7 (Day 36) for a total of 7 weeks
Population: Safety Population: safety population is defined as all subjects who received at least 1 dose of study drug and had at least one post-baseline safety assessment.
Measure: Mean (Standard Deviation); unit: percent change in IA behaviors
Arm/Group | Placebo | Flexible Dose of SPN-810
Number analyzed (Participants) | 20 | 21
percent change in IA behaviors | -31.73 (25.510) | -35.66 (77.422)

2. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression (IA) Measured by Clinical Global Impression - Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of the severity of IA behaviors. CGI-S was evaluated by the Investigator at each visit on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill.
  Data represent the change between Baseline (Visit 3/Day 1) and four time points: Visit 4 (Day 15); Visit 5 (Day 22), Visit 6 (Day 29) and Visit 7 (Day 36).
Time Frame: From Baseline/Visit 3 (Day 1) to Visit 4 (Day 15), Visit 5 (Day 22), Visit 6 (Day 29), Visit 7 (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Flexible Dose of SPN-810
Number analyzed (Participants) | 20 | 21
score on a scale
  Visit 4: number analyzed (Participants) | 19 | 19
  Visit 4 | -0.5 (0.77) | -0.6 (0.69)
  Visit 5: number analyzed (Participants) | 19 | 18
  Visit 5 | -0.7 (0.73) | -1.1 (0.94)
  Visit 6: number analyzed (Participants) | 18 | 17
  Visit 6 | -1.1 (0.96) | -1.2 (0.90)
  Visit 7: number analyzed (Participants) | 18 | 17
  Visit 7 | -1.3 (1.03) | -1.4 (1.00)

3. Secondary Outcome: Effect of SPN810 on Retrospective-Modified Overt Aggression Scale (R-MOAS) Total Score
Description: R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (VE, PH, PR, SE). For each open question in each area, the parent-rated the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: Verbal Incidents (VE)=1, Incidents Toward Other (PH)=4, Incidents Involving Property (PR)=2 and Incidents Directed Toward Self (SE)=3. Therefore, the sum of each area yields a maximum weighted score of 20 (VE), 120 (PH), 60 (PR), and 90 (SE). The total score is the sum of the four area scores or 0-290; the higher the score, the more severe the aggressive behavior is.
  Data represent the total score change between the Baseline (Visit 3/Day 1) and four time points: Visit 4 (Day 15); Visit 5 (Day 22), Visit 6 (Day 29), and Visit 7 (Day 36).
Time Frame: From Baseline/Visit 3 (Day 1) to Visit 4 (Day 15), Visit 5 (Day 22), Visit 6 (Day 29) and Visit 7 (Day 36).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Flexible Dose of SPN-810
Number analyzed (Participants) | 20 | 21
units on a scale
  VE Score Visit 4: number analyzed (Participants) | 19 | 19
  VE Score Visit 4 | -1.4 (3.89) | -5.9 (4.32)
  PH Score Visit 4: number analyzed (Participants) | 19 | 19
  PH Score Visit 4 | -3.4 (9.55) | -4.8 (12.62)
  PR Score Visit 4: number analyzed (Participants) | 19 | 19
  PR Score Visit 4 | -2.4 (7.62) | -6.6 (6.57)
  SE Score Visit 4: number analyzed (Participants) | 19 | 19
  SE Score Visit 4 | -1.9 (6.94) | -4.6 (10.46)
  Total Score Visit 4: number analyzed (Participants) | 19 | 19
  Total Score Visit 4 | -9.1 (16.53) | -21.9 (19.22)
  VE Score Visit 5: number analyzed (Participants) | 19 | 18
  VE Score Visit 5 | -3.7 (3.93) | -7.3 (5.03)
  PH Score Visit 5: number analyzed (Participants) | 19 | 18
  PH Score Visit 5 | -8.6 (8.87) | -12.4 (12.34)
  PR Score Visit 5: number analyzed (Participants) | 19 | 18
  PR Score Visit 5 | -5.4 (9.93) | -9.1 (8.41)
  SE Score Visit 5: number analyzed (Participants) | 19 | 18
  SE Score Visit 5 | -2.1 (7.88) | -6.0 (9.09)
  Total Score Visit 5: number analyzed (Participants) | 19 | 18
  Total Score Visit 5 | -19.8 (23.37) | -34.9 (25.76)
  VE Score Visit 6: number analyzed (Participants) | 18 | 17
  VE Score Visit 6 | -5.4 (4.17) | -6.6 (5.12)
  PH Score Visit 6: number analyzed (Participants) | 18 | 17
  PH Score Visit 6 | -7.8 (17.91) | -12.2 (11.00)
  PR Score Visit 6: number analyzed (Participants) | 18 | 17
  PR Score Visit 6 | -7.3 (9.38) | -7.6 (6.13)
  SE Score Visit 6: number analyzed (Participants) | 18 | 17
  SE Score Visit 6 | -3.2 (7.94) | -3.5 (6.30)
  Total Score Visit 6: number analyzed (Participants) | 18 | 17
  Total Score Visit 6 | -23.7 (32.21) | -30.0 (15.41)
  VE Score Visit 7: number analyzed (Participants) | 18 | 17
  VE Score Visit 7 | -5.7 (4.31) | -7.5 (4.99)
  PH Score Visit 7: number analyzed (Participants) | 18 | 17
  PH Score Visit 7 | -12.9 (13.89) | -11.3 (9.51)
  PR Score Visit 7: number analyzed (Participants) | 18 | 17
  PR Score Visit 7 | -8.3 (8.85) | -9.6 (6.60)
  SE Score Visit 7: number analyzed (Participants) | 18 | 17
  SE Score Visit 7 | -3.3 (9.14) | -3.9 (6.85)
  Total Score Visit 7: number analyzed (Participants) | 18 | 17
  Total Score Visit 7 | -30.2 (29.99) | -32.3 (15.45)

4. Secondary Outcome: Effect of SPN-810 on Retrospective-Modified Overt Aggression Scale (R-MOAS) Remission Rate
Description: The treatment effect on the R-MOAS was assessed to capture the severity of the aggressive behaviors. The remission rate was defined as percentage of subjects with a R-MOAS total score ≤ 10.
  Data represent the percentage of subjects at four time points during the treatment period: Visit 4 (Day 15); Visit 5 (Day 22), Visit 6 (Day 29) and Visit 7 (Day 36).
Time Frame: Visit 4 (Day 15), Visit 5 (Day 22), Visit 6 (Day 29) and Visit 7 (Day 36)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Flexible Dose of SPN-810
Number analyzed (Participants) | 20 | 21
percentage of participants
  Visit 4: number analyzed (Participants) | 19 | 19
  Visit 4 | 10.5 | 26.3
  Visit 5: number analyzed (Participants) | 19 | 18
  Visit 5 | 21.1 | 33.3
  Visit 6: number analyzed (Participants) | 18 | 17
  Visit 6 | 27.8 | 41.2
  Visit 7: number analyzed (Participants) | 18 | 17
  Visit 7 | 38.9 | 58.8

ADVERSE EVENTS:
Time Frame: Baseline/Visit 3 (Day 1) to Visit 8 (Day 46)-End of Study, a total of 46 days
Description: Adverse events reporting pertains to the Safety Population, defined as all subjects who received at least 1 dose of study drug and had at least one post-baseline safety assessment
Arm/Group | Placebo | Flexible Dose of SPN-810
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 8/20 | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Flexible Dose of SPN-810 (N=21)
Headache (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 2 | 0
Dystonia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03597503/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT03597503/SAP_001.pdf